CLINICAL TRIAL: NCT05640024
Title: Prospective Cohort Study for Validation of Predictive Immune Biomarkers of Response to PAPR Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1170
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA based on whole blood. The investigator will peripheral blood from ovarian cancer patients receiving PARP inhibitor for every three months until progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increasing number of ovarian cancer patients are receiving PARP inhibitor as maintenance therapy. Predictive factors to PARP inhibitor other than BRCA mutation or HRD status are unknown. Previous study, we analyzed the dynamic immunological changes in peripheral T cells during PARP inhibitor maintenance therapy and found predictive biomarkers. The purpose of this study is to prospectively validate the biomarkers for predicting response to PAPR inhibitors in ovarian cancer. We collect serial blood samples (before initiation of therapy and after 1, 3, and 6 months) in ovarian cancer patients who receive PARP inhibitor and analyze immunological characteristics of peripheral CD8 and regulatory T cells. Through assessment of the baseline properties and dynamic changes in T cells, we aim to validate the predictive biomarker and develope promising novel targets to enhancing survival outcomes of high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of epithelial ovarian cancer, 2. Presence of germline or somatic BRCA mutational status result, 3. Advanced or recurrent ovarian cancer patients who responded to their most recent platinum-based chemotherapy and plan to start PARPi (olaparib or niraparib) maintenance therapy.

Exclusion Criteria:

1. Patients who refuse to participate, 2. Patients having difficulty understanding the protocol due to language barrier

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients who receive PARP inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Validation of biomarkers for predicting response to PAPR inhibitor | The primary endpont will be accessed 12 months after last patient registration.
  Investigators will utilize baseline peripherap blood mononuclear cells (PBMCs) to validate predictive biomarkers to PARP inhibitor. Response to PAPR inhibitor was defined by BRCA1/2 status and duration of PAPR inhibitor treatment.

SECONDARY OUTCOMES:
Identify dynamic immunological changes during PAPR inhibitor therapy | Immunological changes (Time Frame: 6 months
  Investigators will utilize serial samples to identify dynamic immunological changes during PAPR inhibitor therapy.
Identify promising novel targets to enhance survivla outcomes of high-risk pateints in PAPR inhibitor therapy. | Identify promising novel targets (Time Frame: 12 months)
  Investigators will utilize serial samples to identify dynamic immunological changes during PAPR inhibitor therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun Lee, Principal Investigator — Yonsei University College of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No